CLINICAL TRIAL: NCT00479362
Title: Randomized Trial of Uninterrupted Versus Interrupted Anticoagulant Therapy in Patients Undergoing Cardiac Pacing Device Implantation
Brief Title: Anticoagulant Therapy During Pacemaker Implantation
Acronym: FINPAC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Turku (Other)
Collaborators: Satakunta Central Hospital (Other); Oulu University Hospital (Other); Tampere University Hospital (Other)
Responsible Party: Principal Investigator, Juhani Airaksinen, Professor, University of Turku
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FINPAC; TAHD-VARF (Former Protocol ID); TV001
Record Dates: First submitted 2007-05-25; First posted 2007-05-28 (Estimated); Last update posted 2012-09-17 (Estimated); Status verified 2012-09

CONDITIONS: Hemorrhage; Thrombosis; Embolism
Keywords: Pacemaker; Cardioverter-defibrillator; Hemorrhage; Hematoma; Thrombosis; Embolism
MeSH Terms: conditions — Hemorrhage; Thrombosis; Embolism; Hematoma | interventions — Warfarin; Aspirin; Defibrillators, Implantable

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 Warfarin Uninterrupted (Experimental): Warfarin therapy is continued without interruption prior to cardiac pacing device implantation
  Interventions: Drug: Warfarin; Device: Permanent pacemaker; Device: Implantable Cardioverter-defibrillator
- 2 Warfarin Interrupted (Active Comparator): Warfarin therapy is discontinued 2 days prior to cardiac pacing device implantation
  Interventions: Drug: Warfarin; Device: Permanent pacemaker; Device: Implantable Cardioverter-defibrillator
- 3 Aspirin Group (Sham Comparator): Patients with aspirin therapy during implantation
  Interventions: Drug: Aspirin; Device: Permanent pacemaker; Device: Implantable Cardioverter-defibrillator
- 4 No Antithrombotic Group (Other): No antithrombotic treatment during operations
  Interventions: Device: Permanent pacemaker; Device: Implantable Cardioverter-defibrillator

INTERVENTIONS:
Drug: Warfarin — Warfarin is either interrupted or uninterrupted prior to device implantation
  Other Names: Marevan, ATC code B01AA03; Marevan Forte, ATC code B01AA03
  Arms: 1 Warfarin Uninterrupted; 2 Warfarin Interrupted
Drug: Aspirin — Aspirin is continued without interruption prior to device implantation
  Other Names: Acethyl Salcylic Acid; Primaspan, ATC code B01AC06; Disperin, ATC code B01AC06; Aspirin Cardio, ATC code B01AC06
  Arms: 3 Aspirin Group
Device: Permanent pacemaker — Devices are implanted tailored each patient's clinical condition and need following local practices, national and international guidelines.
  Other Names: Pacing Device Implantation
Device: Implantable Cardioverter-defibrillator — Devices are implanted tailored each patient's clinical condition and need following local practices, national and international guidelines.
  Other Names: ICD

SUMMARY:
There are no established guidelines regarding interruption of warfarin anticoagulant therapy prior to surgical implantation of cardiac pacemakers. Continuing the anticoagulant could potentially result in increased bleeding complications from the implantation surgery, whereas discontinuing the anticoagulant could predispose the patient to blood clots and strokes. In this study we intend to randomly assign warfarin-treated patients either into interrupted or continued warfarin therapy prior to pacemaker implantation with the purpose of establishing the rate of complication in these groups. Our hypothesis is that a cardiac pacing device can be safely implanted without discontinuation of the anticoagulant therapy.

DETAILED DESCRIPTION:
Despite greatly increased utilization of pacemaker and internal cardioverter-defibrillator (ICD) therapy for various indications in recent years, there are relatively few published studies on bleeding complications associated with the implantation of these devices. The purpose of our study is to assess the incidence and severity of hemorrhagic complications resulting from pacemaker and ICD implantation in patients treated with oral anticoagulant warfarin or acetyl salicylic acid.

There are no unified guidelines regarding warfarin use during pacemaker implantation. A case by case approach is commonly employed regarding whether to interrupt or to continue anticoagulant therapy prior to the procedure. Interrupting the therapy may expose the patient to thromboembolic complications, whereas continuing it can increase the risk of perioperative bleeding. Thus, either approach could potentially increase patient morbidity and prolong the hospital stay. Therefore, an evidence based choice of an appropriate approach in preparing the anticoagulant-treated patients for pacemaker implantation could have significant impact on both patient safety and over-all procedural cost.

We intend to assess the rate of hemorrhagic and thrombotic complications as well as the length of hospital stay associated with pacemaker or ICD implantation in patients randomized either to continue or to interrupt their warfarin treatment. One control group will be formed of pacemaker-receiving patients on acetyl salicylic acid as well as one group of patients on no medications affecting the coagulation system or thrombocyte aggregation. Potential risk factors for bleeding or thromboembolic complications will be searched.

A total of 400 patients will be recruited into this multicenter study conducted at five hospitals in Finland. Warfarin users (n=200) will be randomly allocated into two groups: A. uninterrupted warfarin therapy maintained at accepted intensity (INR 2 to 3), and B. interruption of warfarin 2 days prior to device implantation. Control groups will comprised as described above with one hundred patients in each. The end-points of the study are: occurrences of major bleeding, haemorrhages and hematomas at pacemaker pocket, utilization of adjunctive therapies to control bleeding (e.g. Vitamin K or Fresh frozen plasma), need for surgical wound revision and thromboembolic complications. The duration of hospital stay will also be recorded. At two of the centres (Turku University Hospital and Satakunta Central Hospital) all patients will also be randomly assigned into two groups in which the implantation procedure will either be or not be guided by venous angiography.

Patients willing to participate in the study will receive both verbal and written information on the study and they will be asked to sign an informed consent. All devices will be implanted in a normal fashion according to generally accepted clinical guidelines. A variety of clinical and laboratory variables will be recorded in each study group to identify risk factors for bleeding and thromboembolism.

The aims of our study are to establish among patients implanted with pacemakers (1) whether uninterrupted warfarin therapy will increase the rate and severity of bleeding complications, (2) whether interruption of warfarin results in increased thromboembolic events, (3) whether aspirin treatment increases bleeding complications compared, and we also seek to identify factors predisposing to haemorrhagic complications.

Our main hypothesis is that a cardiac pacing device can be safely implanted without discontinuation of the anticoagulant therapy.

ELIGIBILITY:
Inclusion Criteria:

* all patients admitted for implantation of a first permanent cardiac pacing device are eligible

Exclusion Criteria:

* known coagulation disorder or bleeding diathesis
* contraindications for pacing device implantation
* mechanical prosthetic heart valve
* other absolute contraindication to interrupt warfarin
* INR (international normalized ratio) above 3.0 2 days prior to implantation
* significant anemia (hemoglobin less than 100 g/L)
* warfarin interrupted before randomization and INR subtherapeutic (below 2.0)
* not to be randomized to venography: contraindications to radiographic contrast dye

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 447 (Actual)
Dates: Start 2005-09; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Measure: rate of haemorrhagic and thromboembolic complications | within first four weeks

CONTACTS AND LOCATIONS:
Overall Officials: Juhani Airaksinen, MD, Study Director — University of Turku, Turku University Hospital; Petri Korkeila, MD, Principal Investigator — Turku University Hospital
Locations (1):
- Turku University Hospital, Turku, Finland